CLINICAL TRIAL: NCT04158817
Title: Gallium-68 Labelled THP-PSMA for the Clinical Stage and Restage of Prostate Cancer Patients
Brief Title: 68Ga-THP-PSMA PET/CT in Prostate Cancer: Clinical Stage and Restage
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: NanoMab Technology (UK) Limited (Industry)
Responsible Party: Principal Investigator, Zhao Jin Hua, MD, Director Department of Nuclear Medicine, Principal Investigator, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: [2018]15
Record Dates: First submitted 2019-10-22; First posted 2019-11-12 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer
Keywords: 68Ga-THP-PSMA; PET/CT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): All Prostate cancer patients recruited to the study will be administered 2.11 MBq/kg of 68Ga-THP-PSMA in a single dose injection.
  Interventions: Drug: 68Ga-Labeled PSMA; Drug: Non-labeled PSMA

INTERVENTIONS:
Drug: 68Ga-Labeled PSMA — All participants in the study will be injected with 68Ga-THP-PSMA at a dose of 2.11 MBq/kg in a single dose injection.
  Other Names: 68Ga-THP-PSMA
Drug: Non-labeled PSMA — Patient will be injected with microdose (<100 ug) of THP-PSMA
  Other Names: THP-PSMA

SUMMARY:
To evaluate the dosimetry, safety and the detection rate of 68Ga-THP-PSMA PET/CT for identifying the site of prostate cancer metastasis and relapse. It is also to evaluate the association of clinical/pathologic features and 68Ga-THP-PSMA PET/CT detection rate and compare 68Ga-THP-PSMA PET/CT with other imaging procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male, age 18 years or older
2. Prior diagnosis of prostatic cancer
3. Willing to participate in this study and given written informed consent
4. AST, ALT, BUN, Cr not more than double the normal values
5. Subjects of childbearing potential must be willing to undergo a pregnancy test prior to enrolment

Exclusion Criteria:

1. Subjects with pacemakers
2. Hepatitis B virus infection (including carriers) at screening, i.e. hepatitis B surface antigen (HBsAg) positive, or hepatitis C antibody (anti-HCV) positive, or acquired immunodeficiency disease (HIV) infected, or serum syphilis positive person
3. Abnormal liver function during baseline screening period: AST or ALT> 2 times the upper limit of normal value (ULN), if the marginal increase of a single index is judged as having no clinical significance by the investigator, it can be retested during the screening period. Once, if more than 2 times ULN after retesting, consider enrolling).
4. Impaired renal function during screening: serum creatinine or urea nitrogen > 1.5 times ULN.
5. Within 4 months prior to the baseline screening period, myocardial infarction or other cardiac events requiring hospitalization (unstable angina, etc.), cerebrovascular accident, transient ischemic attack, acute congestive Heart failure or severe arrhythmia (ventricular arrhythmia, atrioventricular block above II)
6. Subjects with pulmonary embolism or deep vein thrombosis
7. Various infections that the investigators consider unsuitable for study, including but not limited to patients with various infections requiring further treatment, such as urinary tract infections, respiratory infections, and diabetic foot infections.
8. Patients with abnormal thyroid function during baseline screening period (including but not limited to active hyperthyroidism, hypothyroidism or Hashimoto's thyroiditis)

Ages: 18 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 8 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
The maximal standard uptake value | 2 years
  The tumor SUVmax of patients will be measured using Region Of Interest.
The measurement of PSA | 2 years
  The PSA level (ng/mL) of patients will be tested by hemanalysis
68Ga-THP-PSMA PET/CT in prostate cancer: clinical stage and restage | 2 years
  Visual analysis will be carried out by 4 experienced nuclear medicine physicians to observe the uptake of 68Ga-THP-PSMA in prostate malignant lesions. A 4 point method will be used to interpret the scans for abnormalities. It is categorized as such: score 0, no abnormal increased uptake; score 1, low increased uptake; score 2, moderate increased uptake; score 3, high increased uptake. The lesion will be considered positive for malignancy if the score is 2 or higher.

SECONDARY OUTCOMES:
The correlation analysis | 2 years
  The IHC results of prostate malignant lesions will be used as golden standard to evaluate the sensitivity and specificity of 68Ga-THP-PSMA PET/CT.
The dosimetry assessment | 2 years
  To evaluate the dosimetry of 68Ga-THP-PSMA, patients (n = 5) will undergo whole-body planar imaging at different time points (10 min, 1 h, 2 h and 3 h after injection) to obtain radiation dosimetry data. A calibration source of 37 MBq at injection time will be placed above the head of each patient to provide quantitative calibration of counts to activity.
The safety evaluation | 2 years
  Drug-related adverse reactions will be recorded during the 7-d follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Jinhua Zhao, PhD, Principal Investigator — Department of Nuclear Medicine, Shanghai General Hospital
Locations (1):
- Shanghai General Hospital, Shanghai, China